CLINICAL TRIAL: NCT02712645
Title: A Multicenter Breast Cancer Biospecimen Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Luminist, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LUM-BC-1.0
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

SUMMARY:
This study is being performed to collect blood for the development of noninvasive tests that can screen for or diagnose cancer. Blood samples will be collected from women who are scheduled to have breast biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Females of all racial and ethnic groups who are 40 years or older.
2. Women must:

   1. have suspected neoplasm of the breast (BIRADS 4 or 5) based on the results of any breast screening or diagnostic imaging, such as mammogram, and
   2. be selected or scheduled for a breast biopsy which has not yet been conducted at the time of enrollment.

Exclusion Criteria:

1. Inability to sign informed consent.
2. More than one radiological finding.
3. Any current or prior cancer (with the exception of non-melanoma skin cancer or a suspected breast malignancy targeted for biopsy).
4. Any known or suspected acute illness or condition - including acute infections - at the time of enrollment or within the previous 30 days.
5. Any surgery, hospitalization, or institutionalization (such as in a nursing home) during the previous 3 months.
6. Received any experimental therapeutic treatment during the previous 3 months.
7. Received any blood product transfusion within the previous 3 months.
8. Use of illegal drugs during the previous 3 months.
9. Pregnant or nursing at the time of enrollment or in the preceding 12 months.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women scheduled for a breast biopsy.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with untreated newly diagnosed breast cancer. | 1 Year

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Redding, California
  - Dallas, Texas